CLINICAL TRIAL: NCT04996212
Title: Study of the Effectiveness of a Cardiorespiratory Telerehabilitation Program in Persistent COVID-19 Patients. Randomized Clinical Trial.
Brief Title: Telerehabilitation Program in Persistent COVID-19
Acronym: COVIDPERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1573778
Record Dates: First submitted 2021-08-05; First posted 2021-08-09 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2021-08

CONDITIONS: Coronavirus Infection; Respiratory Disease
Keywords: Covid-19; Physical Therapy; Dyspnea; Fatigue; Online Health; Functional Status
MeSH Terms: conditions — Coronavirus Infections; Respiration Disorders; COVID-19; Dyspnea; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking APP Group (Experimental)
  Interventions: Procedure: Walking APP Group
- Functional APP Group (Experimental)
  Interventions: Procedure: Functional APP group

INTERVENTIONS:
Procedure: Walking APP Group — The participants of this group will be explained their treatment plan by a physiotherapist who will contact them through a video call. This treatment will consist of breathing exercises (abdominodiaphragmatic and pursed lips breathing) and 3 days of aerobic exercise: walking.
  Participants will consult their treatment plan through an application that will be installed on their mobile phone. They will start with 25 minutes of walking and will increase progressively until they reach 45 minutes.
  A biweekly follow-up will be carried out through a phone call by the research team to find out their health status and evolution with the assigned treatment.
  Participants must perform the proposed exercises, 5 days a week, once a day In addition to the respiratory physiotherapy guideline, they will be given the health education manual.
  Arms: Walking APP Group
Procedure: Functional APP group — The participants of this group will be explained their treatment regimen by a physiotherapist who will contact them through a video call. This treatment planwill consist of breathing exercises (abdominodiaphragmatic and pursed lips breathing) and 3 days of functional exercise which involve the activation and performance of large muscle groups. Participants will consult their treatment plan through an application that will be installed on their mobile phone.
  A biweekly follow-up will be carried out through a phone call by the research team to find out their health status and evolution with the assigned treatment.
  Arms: Functional APP Group

SUMMARY:
The syndrome characterized by the persistence of symptoms typical of COVID-19, beyond 4 weeks after discharge, is called long COVID. Long COVID affects a high percentage of patients who have suffered from COVID-19, regardless of its severity. The various symptoms present in that patients affect the functionality and physical, mental and psychological capacities of patients. Therefore, it is necessary to implement therapeutic programs, based on exercises and techniques of physiotherapy, to help affected people to resume their work, family, social and sports activities; prior to illness. Given the context in which these programs must be developed, telecare is positioned as the most recommended care method to carry out the rehabilitation of these patients. The general objective of this study is to evaluate the effectiveness of a cardiorespiratory tele-rehabilitation program in persistent COVID-19 patients. Study participants (n=60) will be randomly assigned to one of two intervention groups. Group 1 will combine breathing exercises with aerobic exercise: walk; and group 2 will perform functional exercises in addition to respiratory physiotherapy with. All participants will be evaluated at the beginning of the intervention, at the end of it.

ELIGIBILITY:
Inclusion Criteria:

* Who have been diagnosed with coronavirus infection (PCR + and / or Antigen Test +).
* Have had a mild form of COVID-19 (absence of symptoms or mild symptoms without signs of viral pneumonia or hypoxia).
* Have overcome such infection; and continue to experience persistent symptoms, including dyspnea, fatigue, and / or functional limitation.

Exclusion Criteria:

* Subjects suffering from other pulmonary or cardiac pathologies and / or diabetes, cancer.
* Individuals who required hospitalization, during the acute stage of infection;
* People who continue to obtain a positive PCR and / or positive Antigen Test;
* Those who have not been discharged by their doctor;
* Subjects who show serious symptoms and / or require medical supervision;
* Individuals with an inability to handle the internet and devices, such as mobile phones, computers or tablets; essential for telecare

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Quality of life (EQ-5D-5L) | It will be evaluated in two moments: Pre intervention: before starting the exercise program Post intervention: after 8 weeks of physiotherapy intervention
  The EQ-5D-3L is a short and simple scale consisting of 2 parts. In the first of the pages, a total of 5 questions allow evaluating five different dimensions: mobility, self-care, habitual activities, pain / discomfort and anxiety / depression. In the second part, through a Visual Analogue Pain Scale (VAS), the patient can quantify, from 0 to 100, her perceived health status at the time of evaluation

SECONDARY OUTCOMES:
Quality of life (EQ-5D-5L) Change from Baseline PostCovid-19 Functional Satatus Scale at five months (PCFSS) | It will be evaluated in two moments: Pre intervention: before starting the exercise program Post intervention: after 8 weeks of physiotherapy intervention
  The PCFS items assess the functional limitations that post-COVID-19 patients The EQ-5D-3L is a short and simple scale consisting of 2 parts. In the first of the pages, a total of 5 questions allow evaluating five different dimensions: mobility, self-care, habitual activities, pain / discomfort and anxiety / depression. In the second part, through a Visual Analogue Pain Scale (VAS), the patient can quantify, from 0 to 100, her perceived health status at the time of evaluation
Fatigue Assessment Scale (FAS) | It will be evaluated in two moments: Pre intervention: before starting the exercise program Post intervention: after 8 weeks of physiotherapy intervention
  The scale consists of 10 items through which the fatigue experienced by the subject can be assessed at two levels: physical and mental.
  Participants in this study must answer how often the situations described in each item on the scale occur. To do this, they must quantify each statement with a number from 1 to 5, where 1 is never; and 5, always.
London Chest Activity of Daily Living Scale (LCADL) | It will be evaluated in two moments: Pre intervention: before starting the exercise program Post intervention: after 8 weeks of physiotherapy intervention
  The LCADL was designed with the purpose of assessing the level of dyspnea, reported by patients with pulmonary pathology, during the performance of ADL. The LCADL scale therefore makes it possible to assess and adequately monitor the functional deterioration that patients experience as a consequence of their dyspnea. Throughout its development, this scale explores 4 different dimensions: self-care, home activities, physical activity and leisure activities.
Hospital Anxiety and Depression Scale (HADS) | It will be evaluated in two moments: Pre intervention: before starting the exercise program Post intervention: after 8 weeks of physiotherapy intervention
  The HADS scale is a widely used instrument to assess the degree of emotional distress suffered by people with pathology. The scale consists of 14 items that consider cognitive, affective and behavioral aspects; but not somatic. The original version of the HADS has been validated and translated into different languages, including Spanish
Perceived Stress Scale (PSS) | It will be evaluated in two moments: Pre intervention: before starting the exercise program Post intervention: after 8 weeks of physiotherapy intervention
  The PSS allows evaluating the level of stress perceived by patients during the last month It is made up of 14 items that explore the thoughts and feelings of the respondent that can be related to high levels of stress. The higher the score, the higher the level of perceived stress.
Beck Depression Inventory (BDI-2) | It will be evaluated in two moments: Pre intervention: before starting the exercise program Post intervention: after 8 weeks of physiotherapy intervention
  The BDI-2, through its 21 items, aims to help the health professional to identify and measure the severity of symptoms, typical of a depressive process, in the adult population
Exercise tolerance. Thirty Seconds Sit-To-Stand | It will be evaluated in two moments: Pre intervention: before starting the exercise program Post intervention: after 8 weeks of physiotherapy intervention
  Exercise tolerance will be assessed using the Thirty Seconds Sit-To-Stand test (30stst), as it has proven to be a useful test to evaluate the strength and endurance of the lower limbs and determine the patient's tolerance to physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Cortés Amador, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
IPD are not to be shared with other researchers